CLINICAL TRIAL: NCT03139760
Title: POWERSforID: Personalized Online Weight and Exercise Response System for Adults With Intellectual Disability
Brief Title: POWERSforID: A Telehealth Weight Management System for Adults With Intellectual Disability
Acronym: POWERSforID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, James Rimmer, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: F141230005
Record Dates: First submitted 2017-04-22; First posted 2017-05-04 (Actual); Last update posted 2018-11-15 (Actual); Status verified 2018-11

CONDITIONS: Intellectual Disability; Weight Loss; Motivational Interviewing; Telehealth
MeSH Terms: conditions — Intellectual Disability; Weight Loss

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- POWERSforID (Experimental): POWERSforID intervention group
  Interventions: Behavioral: POWERSforID
- Control (No Intervention): Usual clinical care

INTERVENTIONS:
Behavioral: POWERSforID — Feasibility and outcomes associated with use of the POWERSforID system and coaching phone calls over the course of 24 weeks
  Arms: POWERSforID

SUMMARY:
POWERSforID is a 24 week randomized control trial designed to assess the feasibility of a telehealth and coaching intervention for improving health outcomes of adults with intellectual disability. Recruitment is conducted through a disability health clinic located in Colorado Springs, CO.

DETAILED DESCRIPTION:
POWERS (Personalized Online Weight and Exercise Response System) platform is a novel, multifocal-centered tailored intervention utilizing an innovative online tool designed to facilitate improvements in physical activity and nutritional behaviors. Aim 1 of this protocol is to customize the POWERS platform, demonstrated effective in previous research, for adults with intellectual disability (ID) and their caregivers to be referred to as POWERSforID. The POWERSforID intervention is designed to achieve weight loss and improve specific health markers while respecting and supporting the needs of the participants with ID as well as their caregivers. Aim 2 of the project is to conduct a pilot study to assess the usability and feasibility of the POWERSforID system and intervention with 5 adults with ID and their caregiver and improve the system based on pilot data. Aim 3 of the protocol is to conduct a randomized controlled trial (RCT) to examine the effect of POWERSforID on educating and coaching caregivers about nutrition and exercise and thus improving health status and reducing body weight in obese adults with ID. The investigators hypothesize that the obese participants in the intervention group (POWERSforID) will evidence significantly greater weight loss and improved health status (i.e. lower waist circumference, blood pressure, decreased body fat percentage, and improved blood lipids) compared to a control group. The investigators also hypothesize that both adults with ID and their caregivers will demonstrate improved knowledge, attitudes, and self-efficacy related to diet and exercise.

ELIGIBILITY:
Inclusion Criteria:

* Participants with intellectual disability (ID) who meet the following inclusion criteria are eligible to participate in the study:

  * Body Mass Index > or equal to 30 kg/m2;
  * Diagnosis of mild or moderate ID;
  * 25 to 50 years of age;
  * Medical provider approval to participate in a weight loss program;
  * Has a caregiver who agrees to participate in the study and provides services 4 days a week or more to the adult with ID;
  * Has access to a computer with internet throughout the week.

Exclusion Criteria:

* Currently on a weight loss program;
* Medical conditions that prevent participation as noted by the medical provider or legal guardian including heart and/or renal disease;
* Behavioral issues determined by the DDHC Behavioral Health staff;
* Unable to walk or exercise due to a mobility impairment or medical condition;
* Judged to have insufficient capacity to consent or assent as assessed using the "Supplemental Consent Document".

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Participation in weekly phone calls | 24 weeks
  Number of weekly intervention phone calls attended or missed
Number of logins to the POWERSforID website | 24 weeks
  Number of times the POWERSforID website is accessed to journal health related behaviors

SECONDARY OUTCOMES:
Weight loss | 24 weeks
  Weight change measured in kilograms

OTHER OUTCOMES:
Physical activity questionnaire | 24 weeks
  The questionnaire includes assessment of perceived barriers to physical activity and physical activity participation.
Mood/Psychosocial questionnaire | 24 weeks
  Measured by the Glasgow depression scale, Psychosocial questionnaire for individuals with ID, scale for perceived physical and nutrition related barriers
Dietary recall questionnaire | 24 weeks
  The questionnaire includes assessment of type of foods consumed.

CONTACTS AND LOCATIONS:
Overall Officials: James Rimmer, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Neumeier WH, Guerra N, Thirumalai M, Geer B, Ervin D, Rimmer JH. POWERS forID: Personalized Online Weight and Exercise Response System for Individuals with Intellectual Disability: study protocol for a randomized controlled trial. Trials. 2017 Oct 23;18(1):487. doi: 10.1186/s13063-017-2239-2. PMID 29058620